CLINICAL TRIAL: NCT06958913
Title: Comparison of Hemodynamic Response and Cardiac Protective Effects of Propofol Versus Dexmedetomidine at Induction of Anesthesia in Cardiac Surgery: a Randomized Controlled Trial
Brief Title: Effect of Dexmedetomidine on Hemodynamics in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Selvinaz Yüksel Tanrıverdi, MD, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PamukkaleUSyüksel-002
Record Dates: First submitted 2025-04-10; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Use of Dexmedetomidine in Cardiac Surgery (CABG, Valve Replacement or Total Aortic Arch Replacement)
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): In group P, 0.125 cc/kg saline infusion was administered in 10 minutes. Fentanyl was administered at a dose of 3 mcg/kg at 5 minutes of this application. Then propofol was administered until the eyelash reflex disappeared and the BIS value was 40. 0.6 mg/kg rocuronium was administered to facilitate intubation. All patients received 8 mg dexamethasone and lidocaine at a dose of 1 mg/kg.
  Interventions: Drug: Propofol group
- Group DP (Experimental): In group DP, dexmedetomidine at a dose of 0.5 mck/kg was administered over 10 minutes. At the 5th minute of this infusion, fentanyl was administered at a dose of 3 mcg/kg. Propofol was added until the BIS value was 40. The patients received 0.6 mg/kg rocuronium, 8 mg dexamethasone, and 1 mg/kg lidocaine.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol group — In group P, 0.125 cc/kg saline infusion was administered in 10 minutes. Fentanyl was administered at a dose of 3 mcg/kg at 5 minutes of this application. Then propofol was administered until the eyelash reflex disappeared and the BIS value was 40. 0.6 mg/kg rocuronium was administered to facilitate intubation. All patients received 8 mg dexamethasone and lidocaine at a dose of 1 mg/kg.
  Arms: Group P
Drug: Dexmedetomidine — In group DP, dexmedetomidine at a dose of 0.5 mck/kg was administered over 10 minutes. At the 5th minute of this infusion, fentanyl was administered at a dose of 3 mcg/kg. Propofol was added until the BIS value was 40. The patients received 0.6 mg/kg rocuronium, 8 mg dexamethasone, and 1 mg/kg lidocaine.
  Arms: Group DP

SUMMARY:
It is important to establish a stable haemodynamics in patients undergoing cardiac surgery. Haemodynamic depression is common during induction of anaesthesia [1]. Sympathetic response due to tracheal intubation creates unwanted hypertensive responses on haemodynamics. Dexmedetomidine decreases stress responses and may provide a stable haemodynamics in situations such as surgery or induction of anaesthesia [2-4]. It may increase the tendency to hypotension and bradycardia by weakening the hyperdynamic response caused by sympathetic effect [5,6]. Concurrent use of dexmedetomidine may reduce anaesthetic opioid doses and provide more stable haemodynamics on systolic arterial pressure in patients undergoing CABG [7].

During cardiopulmonary bypass, dexmedetomidine may provide myocardial protection by exerting anti-inflammatory effects and may be beneficial for rapid recovery [6,8,9]. In cardiac surgery, dexmedetomidine provided bidirectional regulation of the anti-inflammatory response in which it showed antioxidant properties by inhibiting proinflammatory cytokine production and lipid peroxidation [10,11]. Dexmedetomidine in combination with propofol resulted in lower myocardial enzyme values than propofol alone [12]. The cardioprotective effects of propofol are dose-dependent; however, haemodynamic instability may be a concern at higher doses. In addition, dexmedetomidine may be considered a valid alternative to propofol, mainly because of its haemodynamic stability and possible myocardial protective effects [13]. It has been shown that dexmedetomidine pretreatment in valvular heart surgery can reduce the dose of propofol and the duration of mechanical ventilation and provide myocardial protection without an increase in adverse events [14]. Our study had two aims. The first was to provide a more stable haemodynamics by adding dexmedetomidine to induction in open cardiovascular surgery anaesthesia. Hypotension during induction and hypertensive response during tracheal intubation were tried to decrease. The second was to evaluate the effect of dexmedetomidine on cardiac enzymes only during induction, i.e. to evaluate its cardiac protective efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who underwent cardiovascular surgery (coronary artery bypass grafting, valve replacement or total aortic arch replacement) for ischaemic heart disease, valvular disease or aortic arch aneurysm were included.

Exclusion Criteria:

* Severe cardiovascular disease [(NYHA class 4 or left ventricular ejection fraction (LVEF) less than 30%)] ,
* Concomitant systemic disorders (e.g. patients with severe liver dysfunction or chronic renal failure on haemodialysis),
* Pregnant women,
* Emergency cases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Effect of dexmedetomidine on systolic blood pressure (SBP mm/hg) | SBP was recorded as the first basal value after monitoring of the patient. Data were recorded at 5 and 10 minutes after the start of induction and just before intubation. The highest value in the first 5 minutes after intubation was recorded.
  Datawere (SBP mm/hg) recorded during induction, before intubation, after intubation and before the start of surgery.
Effect of dexmedetomidine on diastolic blood pressure (DBP mm/hg) | DBP was recorded as the first basal value after monitoring of the patient. Data were recorded at 5 and 10 minutes after the start of induction and just before intubation. The highest value in the first 5 minutes after intubation was recorded.
  Datawere(DBP mm/hg) recorded during induction, before intubation, after intubation and before the start of surgery.
Effect of dexmedetomidine on heart rate (HR bpm) | HR was recorded as the first basal value after monitoring of the patient. Data were recorded at 5 and 10 minutes after the start of induction and just before intubation. The highest value in the first 5 minutes after intubation was recorded.
  Datawere (HR bpm) recorded during induction, before intubation, after intubation and before the start of surgery.
Effect of dexmedetomidine on mean arterial pressure (MAP mm/hg) | MAP was recorded as the first basal value after monitoring of the patient. Data were recorded at 5 and 10 minutes after the start of induction and just before intubation. The highest value in the first 5 minutes after intubation was recorded.
  Datawere (MAP mm/hg) recorded during induction, before intubation, after intubation and before the start of surgery.

SECONDARY OUTCOMES:
Creatin kinase MB (IU/L) level for cardiac protective effect | Creatin kinase MB was recorded 1 day before, 1 hour and 24 hours after surgery.
  To evaluate the cardiac protective efficacy of dexmedetomidine, cardiac enzyme CKMB (IU/L) was recorded preoperatively, postoperative 1st hour and 24th hour.
Troponin I (ng/mL) level for cardiac protective effect | Troponin I was recorded 1 day before, 1 hour and 24 hours after surgery.
  To evaluate the cardiac protective efficacy of dexmedetomidine, cardiac enzyme Troponin I (ng/mL) was recorded preoperatively, postoperative 1st hour and 24th hour.

CONTACTS AND LOCATIONS:
Overall Officials: Selvinaz Yüksel Tanrıverdi, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soliman R, Zohry G. The myocardial protective effect of dexmedetomidine in high-risk patients undergoing aortic vascular surgery. Ann Card Anaesth. 2016 Oct-Dec;19(4):606-613. doi: 10.4103/0971-9784.191570. PMID 27716690
- [Background] Kunisawa T, Ueno M, Kurosawa A, Nagashima M, Hayashi D, Sasakawa T, Suzuki A, Takahata O, Iwasaki H. Dexmedetomidine can stabilize hemodynamics and spare anesthetics before cardiopulmonary bypass. J Anesth. 2011 Dec;25(6):818-22. doi: 10.1007/s00540-011-1215-3. Epub 2011 Sep 8. PMID 21901330